CLINICAL TRIAL: NCT06896708
Title: Coronary Computed Tomography Study to Assess the Effect of Intensive Lipid-Lowering Therapy on Coronary Atherosclerotic Plaque Progression in Young and Middle-Aged Patients With Chronic Coronary Syndrome: A Nationwide, Multicentre, Randomized Controlled Trial
Brief Title: Effect of Intensive Lipid-Lowering Therapy on Coronary Atherosclerotic Plaque Progression in Young and Middle-Aged Patients With Chronic Coronary Syndrome
Acronym: CAPITAL-PLAQUE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liu yong (Other)
Responsible Party: Sponsor-Investigator, Liu yong, MD, Guangdong Provincial People's Hospital
Organization: Guangdong Provincial People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2025-394-02
Record Dates: First submitted 2025-02-11; First posted 2025-03-26 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-03

CONDITIONS: Chronic Coronary Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive lipid-lowering strategy (Experimental): LDL-C reduce to <1.0mmol/L and by ≥50% relative to baseline levels.
  Interventions: Drug: Intensive lipid-lowering strategy
- Standard lipid-lowering strategy (Active Comparator): LDL-C reduce to <1.8mmol/L and by ≥50% relative to baseline levels.
  Interventions: Drug: Standard lipid-lowering strategy

INTERVENTIONS:
Drug: Intensive lipid-lowering strategy — The initial recommended therapy is 20mg atorvastatin/10mg rosuvastatin plus Ezetimibe or PCSK9i, and the type and dosage of drugs can be adjusted according to the situation. If the target LDL-C level is not achieved during the Follow-up periods, adjustment of drug type and dosage will be carried out according to procedures defined in the protocol.
  Arms: Intensive lipid-lowering strategy
Drug: Standard lipid-lowering strategy — The initial recommended therapy is 20mg atorvastatin/10mg rosuvastatin, and the type and dosage of drugs can be adjusted according to the situation. If the target L-DLC level is not achieved during the Follow-up periods, adjustment of drug type and dosage will be carried out according to procedures defined in the protocol.
  Arms: Standard lipid-lowering strategy

SUMMARY:
This is a multicenter, open-label, parallel-group, randomized trial to determine if intensive lipid-lowering therapy (goal for LDL-C <1.0 mmol/L and ≥50% reduction frome baseline) could delay progression of coronary atherosclerotic obstructive leisions compared with guideline recommended lipid-lowering therapy (goal for LDL-C <1.8 mmol/L and ≥50% reduction frome baseline) among participants between 18-60 years old with non-invasively managed chronic coronary syndrome (at least one lesion with a 50%-70% stenosis).

DETAILED DESCRIPTION:
Coronary artery disease (CAD) remains the leading cause of mortality worldwide, driven predominantly by the intricate dynamics between lipid metabolism and atherosclerosis. In recent years, the incidence of CAD among middle-aged and young patients has been increasing rapidly, with high-risk of recurrent cardiovascular adverse events. Inadequate lipid control is a significant contributing factor to the progession of CAD. 2024 ESC Guidelines for the managementof chronic coronary syndromes (CCS) and 2024 Chinese guidelines for the diagnosis and management of patients with chronic coronary syndrome highlight the importance of moderate-intensity lipid-lowering therapy control for patients with CCS, goal for LDL-C <1.4 mmol/L or 1.8mmol/L, respectively, and ≥50% reduction frome baseline. The Progression of Early Subclinical Atherosclerosis (PESA) study showed that among individuals with subclinical atherosclerotic plaques, the proportion of plaque regression was highest in young and middle-aged patients, and lower LDL-C levels significantly increased the likelihood of plaque regression. However, for young and middle-aged patients with chronic coronary syndrome, there remains a lack of definitive research data on the effects of intensive lipid-lowering therapy on coronary plaque progession.

CCTA-based noninvasive methods can accurately and sensitively identify and quantify coronary plaque characteristics, providing detailed information about plaque composition, volume, and morphology. This advanced imaging technology allows for precise assessment of high-risk plaque features, such as positive remodeling, low-attenuation plaques, and spotty calcifications, which are critical for evaluating the risk of future adverse cardiovascular events. Additionally, CCTA offers the advantage of longitudinal monitoring, enabling the evaluation of plaque progression or regression in response to lipid-lowering therapy.

This prospective, randomized, open-label, blinded endpoint trial will randomize about 766 participantis aged between 18 and 60 years with with non-invasively managed chronic coronary syndrome (at least one lesion with a 50%-70% stenosis) into the intervention group (goal for LDL-C <1.0 mmol/ and ≥50% reduction frome baseline) and the control group (goal for LDL-C <1.8 mmol/L and ≥50% reduction frome baseline). The aim of this study is to assess the role of intensive lipid-lowering control in delaying plaque progression, especially non-calcified plaques identified by CCTA.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-60 years at screening 2. Stable angina symptoms with suspected or confirmed coronary artery disease; 2. CCTA examination demonstrating: at least one major coronary artery with a diameter of ≥1.5mm that has not been intervened and at least one leision with 50%-70% stenosis.

3. Subjects who have been using statin therapy alone for at least 4 weeks prior to enrollment with a baseline LDL-C ≥1.8mmol/L or subjects who have not initiated lipid-lowering therapy prior to enrollment with a baseline LDL-C≥2.6mmol/L.

Exclusion Criteria:

1. Left main coronary artery disease or severe three-vessel disease;
2. Ultra-high-risk ASCVD patients: ≥2 severe ASCVD events or 1 severe ASCVD event with ≥2 high-risk factors;
3. Use of PCSK9 inhibitors or ezetimibe within 8 weeks prior to study enrollment;
4. The baseline LDL-C was relatively high (LDL-C≥2.6 mmol/L in those taking statins and ≥4.9 mmol/L in those not taking statins).
5. Familial hypercholesterolemia;
6. Known allergy/intolerance to lipid-lowering drugs used in the trial;
7. Patients with severe congestive heart failure, liver or kidney dysfunction, or malignancy;
8. Pregnant or breastfeeding female patients.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 766 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
The composite events of atherosclerotic plaque progression | 12 months
  A composite end-point comprised of plaque progression, nonfatal myocardial infarction, death, or unstable angina driven rehospitalization or revascularization. Plaque progression is defined as an anual progression of PAV measured by CCTA more than 1%. PAV = (total plaque volume/vessel volume) *100%.

SECONDARY OUTCOMES:
Major adverse cardiac events | 12 months
  Composite of nonfatal myocardial infarction, death, or unstable angina driven rehospitalization or revascularization.
Plaque progression event | 12 months
  The proportion of annual change in PAV >1%
Agatston score changes of coronary artery and aortic valve | 12 months
  Evaluating intensive group compared to standard group in Agatston score changes of coronary artery and aortic valve evaluated by CCTA
Percentage change in total coronary atheroma volume | 12 months
  Evaluating intensive group compared to standard group in total atheroma volume change evaluated by CCTA. PAV = (total plaque volume/vessel volume) *100%.
Change in non-obstructive lesion reversal rate | 12 months
  Evaluating intensive group compared to standard group in anual change of rate of improvement from coronary artery obstructive lesions (stenosis rate ≥50%) to non-obstructive lesions (stenosis rate <50%)
Change in total atheroma volume by CCTA | 12 months
  Evaluating intensive group compared to standard group in total atheroma volume change evaluated by CCTA.
Change in total volume and percentage of non-calcified plaques and calcified plaques | 12 months
  Evaluating intensive group compared to standard group in total volume and percentage of non-calcified plaques and calcified plaques' change evaluated by CCTA.
Change in the proportion of high-risk plaques | 12 months
  Evaluating intensive group compared to standard group in the proportion of high-risk plaques' change evaluated by CCTA.
Change in CT Fractional Flow Reserve (CT-FFR) | 12 months
  Evaluating intensive group compared to standard group in CT-FFR change evaluated by CCTA.
Change in perivascular fat attenuation index (FAI) | 12 months
  Evaluating intensive group compared to standard group in FAI change evaluated by CCTA.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Ninth Clinical Medical College of Guangzhou University of Chinese Medicine, Dongguan, Guangdong
  - The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The Eighth Affiliated Hospital of Sun Yat-sen University, Shenzhen, Guangdong
  - Zhongshan People's Hospital, Zhongshan, Guangdong
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mendieta G, Pocock S, Mass V, Moreno A, Owen R, Garcia-Lunar I, Lopez-Melgar B, Fuster JJ, Andres V, Perez-Herreras C, Bueno H, Fernandez-Ortiz A, Sanchez-Gonzalez J, Garcia-Alvarez A, Ibanez B, Fuster V. Determinants of Progression and Regression of Subclinical Atherosclerosis Over 6 Years. J Am Coll Cardiol. 2023 Nov 28;82(22):2069-2083. doi: 10.1016/j.jacc.2023.09.814. PMID 37993199
- [Result] Vrints C, Andreotti F, Koskinas KC, Rossello X, Adamo M, Ainslie J, Banning AP, Budaj A, Buechel RR, Chiariello GA, Chieffo A, Christodorescu RM, Deaton C, Doenst T, Jones HW, Kunadian V, Mehilli J, Milojevic M, Piek JJ, Pugliese F, Rubboli A, Semb AG, Senior R, Ten Berg JM, Van Belle E, Van Craenenbroeck EM, Vidal-Perez R, Winther S; ESC Scientific Document Group. 2024 ESC Guidelines for the management of chronic coronary syndromes. Eur Heart J. 2024 Sep 29;45(36):3415-3537. doi: 10.1093/eurheartj/ehae177. No abstract available. PMID 39210710
- [Result] Raber L, Ueki Y, Otsuka T, Losdat S, Haner JD, Lonborg J, Fahrni G, Iglesias JF, van Geuns RJ, Ondracek AS, Radu Juul Jensen MD, Zanchin C, Stortecky S, Spirk D, Siontis GCM, Saleh L, Matter CM, Daemen J, Mach F, Heg D, Windecker S, Engstrom T, Lang IM, Koskinas KC; PACMAN-AMI collaborators. Effect of Alirocumab Added to High-Intensity Statin Therapy on Coronary Atherosclerosis in Patients With Acute Myocardial Infarction: The PACMAN-AMI Randomized Clinical Trial. JAMA. 2022 May 10;327(18):1771-1781. doi: 10.1001/jama.2022.5218. PMID 35368058
- [Result] Mensah GA, Fuster V, Murray CJL, Roth GA; Global Burden of Cardiovascular Diseases and Risks Collaborators. Global Burden of Cardiovascular Diseases and Risks, 1990-2022. J Am Coll Cardiol. 2023 Dec 19;82(25):2350-2473. doi: 10.1016/j.jacc.2023.11.007. No abstract available. PMID 38092509